CLINICAL TRIAL: NCT03680560
Title: A Phase 1 Study of an Autologous ACTR T Cell Product in Combination With Trastuzumab, a Monoclonal Antibody, in Subjects With HER2-Positive Advanced Malignancies
Brief Title: Study of ACTR T Cell Product in Combination With Trastuzumab in Subjects With HER2-Positive Advanced Solid Tumor Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATTCK-34-01
Record Dates: First submitted 2018-09-14; First posted 2018-09-21 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumor; HER-2 Protein Overexpression
Keywords: HER2; ACTR; ACTR087; ACTR707; T cell; T cell product; adoptive T cells; gene therapy; breast cancer; gastric cancer; gastro esophageal cancer; immunotherapy; solid tumor; adenoid cystic carcinoma
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Carcinoma, Adenoid Cystic | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACTR T cell product in combination with trastuzumab (Experimental)
  Interventions: Biological: ACTR T Cell Product; Drug: Trastuzumab

INTERVENTIONS:
Biological: ACTR T Cell Product — Autologous Antibody-Coupled T Cell Receptor (ACTR) T Cell Product (ACTR707 or ACTR087)
Drug: Trastuzumab — monoclonal antibody targeting HER2

SUMMARY:
This is a Phase 1, open-label, multi-center study to assess safety and determine the recommended phase 2 dose (RP2D) of ACTR T cell product (ACTR707 or ACTR087) in combination with trastuzumab, following lymphodepleting chemotherapy in subjects with HER2-positive advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to study procedures
* Histologically-confirmed Her2 positive advanced solid tumor malignancy with documented disease progression during or immediately following the immediate prior therapy, or within 6 months of completing adjuvant therapy for subjects with breast cancer
* Subjects must have previously received adequate standard therapy for treatment of their malignancy

  * For those with metastatic breast cancer, must have received HER2-directed therapy including trastuzumab, pertuzumab and ado-trastuzumab in any breast cancer disease setting
  * For those with advanced gastric cancer, adequate prior treatment with HER2-directed chemotherapy is required
* At least 1 measurable lesion by iRECIST
* Able to provide fresh tumor biopsy or archived block specimen taken since time of most recent anti-HER2 mAb-directed therapy
* ECOG of 0 or 1
* Life expectancy ≥ 6 months
* LVEF ≥ 50% by MUGA or ECHO
* Absolute neutrophil (ANC) count ≥ 1500/ µL
* Platelet count ≥ 100,000/µL
* Hemoglobin ≥ 9g/dL
* Estimated GFR >30mL/min/1.73m2

Exclusion Criteria:

* glioblastoma multiforme or other primary CNS tumors are excluded
* clinically significant cardiac disease
* clinically significant active infection
* clinical history, prior diagnosis, or overt evidence of autoimmune disease
* current use of more than 5mg/day of prednisone (or an equivalent glucocorticoid)
* Prior treatment as follows:

  * prior cumulative doxorubicin dose greater than or equal to 300 mg/m^2 or equivalent
  * chemotherapy within 2 weeks of enrollment
  * external beam radiation within 2 weeks of enrollment (28 days if CNS-directed therapy)
  * any monoclonal antibody (mAb) or other protein therapeutic containing Fc-domains within 4 weeks of enrollment
  * pertuzumab within 4 months of enrollment
  * Experimental agents within 3 half-lives or 28 days prior to enrollment, whichever is shorter
  * allogeneic hematopoietic stem cell transplant (HSCT)
  * prior infusion of a genetically modified therapy
* Pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ACTR T cell product with trastuzumab as assessed by committee review of dose limiting toxicities (DLTs), incidence and severity of adverse events (AEs) and clinically significant abnormalities of laboratory values | 42 days
Determination of recommended phase 2 dose (RP2D) regimen | 42 days
  Review of DLTs, maximum tolerated dose (MTD), incidence and severity of AEs and clinically significant abnormalities of laboratory values

SECONDARY OUTCOMES:
Anti-tumor activity as measured by overall response rate (ORR) per iRECIST | 52 weeks
Anti-tumor activity as measured best overall response (BOR) | 52 weeks
Anti-tumor activity as measured by duration of response (DOR) | 52 weeks
Anti-tumor activity as measured by progression-free survival (PFS) | 52 weeks
Anti-tumor activity as measured by overall survival (OS) | 52 weeks
Assessment of persistence of ACTR as measured by flow cytometry | 52 weeks
Assessment of persistence of ACTR as measured by quantitative polymerase chain reaction (qPCR) | 52 weeks
Assessment of ACTR phenotype and function as measured by flow cytometry | 52 weeks
Assessment of induction of inflammatory markers and cytokines/chemokines after ACTR T cell product administration | 52 weeks
  Levels of inflammatory markers, cytokines/chemokines in blood
Trastuzumab pharmacokinetics (PK) | 52 weeks
  trastuzumab serum concentration, Area Under the Curve (AUC), trough levels

CONTACTS AND LOCATIONS:
Overall Officials: Glen Weiss, MD, Study Director — Cogent Biosciences, Inc.
Locations (6):
- United States (6):
  - Yale Smilow Cancer Hospital, New Haven, Connecticut
  - Miami University Cancer Center, Miami, Florida
  - The Ohio State University, Columbus, Ohio
  - Sarah Cannon Research Institute/Tennessee Oncology, PLLC, Nashville, Tennessee
  - Baylor Scott & White Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Sponsor Website — https://www.unumrx.com/